CLINICAL TRIAL: NCT05279027
Title: Zirconium Zr 89 Crefmirlimab Berdoxam (Anti-CD8 Minibody) PET/CT Imaging as a Measure of Response in Patients With Advanced Melanoma on Immunotherapy Plus Hydroxychloroquine.
Brief Title: Zr89 + PET Companion Trial
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: ImaginAb, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09620
Record Dates: First submitted 2022-03-08; First posted 2022-03-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Melanoma (Skin)
Keywords: Positron Emission Tomography
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PET imaging (Experimental): This is a single institution, prospective cohort study of 89Zr-Df-IAB22M2C PET/CT as an early measure of response in patients with melanoma.
  Interventions: Drug: Zirconium Zr 89 Crefmirlimab Berdoxa

INTERVENTIONS:
Drug: Zirconium Zr 89 Crefmirlimab Berdoxa — Zirconium Zr 89 Crefmirlimab Berdoxa PET/CT scans pre and post therapy initiation

SUMMARY:
Study of Zirconium Zr 89 Crefmirlimab Berdoxa PET/CT as an imaging biomarker for assessing an early response to therapy in patients with advanced melanoma on immunotherapy and hydroxychloroquine. This study is a companion study to the "LIMIT Melanoma Trial." Patients with melanoma who are potentially eligible for the LIMIT Melanoma Trial and have at least one site of measurable disease based on RECIST 1.1 are potentially eligible. Associations with progression-free survival (PFS) and overall survival (OS) will be tested.

DETAILED DESCRIPTION:
This is a single institution, prospective cohort study of Zirconium Zr 89 Crefmirlimab Berdoxa PET/CT as an early measure of response in patients with melanoma. This study is a companion imaging study to the "LIMIT Melanoma Trial". Patients with melanoma who are candidates for the LIMIT Melanoma treatment trial and are at least 18 years of age may be eligible. All participants will be receiving care at the clinical practices of the University of Pennsylvania. Patients will be approached about study participation regardless of race or ethnic background. We anticipate enrolling up to 20 evaluable participants with melanoma who meet eligibility requirements for this study. An evaluable patient has completed Baseline and at the post-Treatment Zirconium Zr 89 Crefmirlimab Berdoxa PET/CT scans. Accrual is estimated to occur over approximately 3 years.

After undergoing screening assessments and verifying eligibility for study participation subjects will be scheduled to undergo a BaselineZirconium Zr 89 Crefmirlimab Berdoxa PET/CT scan prior to starting immunotherapy + HCQ therapy. For the Baseline study, subjects will be injected with Zirconium Zr 89 Crefmirlimab Berdoxa up to 8 days prior to starting therapy (Day -8 to 0), and will undergo PET/CT imaging 24 ± 4 hours post injection, and prior to therapy administration. Subjects will then undergo a Post-Treatment Zirconium Zr 89 Crefmirlimab Berdoxa PET/CT scan at day 14 (± 4 days) post therapy, which will require administration of Zirconium Zr 89 Crefmirlimab Berdoxa on the day prior to the scan. Zirconium Zr 89 Crefmirlimab Berdoxa PET/CT scans will be acquired with an interval of ≥ 10 days between scans, to ensure that the signal from the previous injection of Zirconium Zr 89 Crefmirlimab Berdoxa has decayed.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, at least 18 years of age
2. History of histologically confirmed melanoma as assessed per medical record review.
3. At least one site of measurable disease (per RECIST 1.1) that is seen on CT, MRI, or FDG PET/CT.
4. Potentially eligible to participate in the LIMIT Melanoma Trial.
5. Patients must have adequate baseline organ function as determined per LIMIT Melanoma Trial (IRB 835033) (these tests will be completed as part of LIMIT trial screening and will not be repeated for the imaging companion study)

   Adequate organ function: per LIMIT Melanoma Trial (IRB 35033)

   System Laboratory Values Hematologic Absolute Neutrophil Count (ANC) ≥ 1.0 x 109/L Hemoglobin ≥ 9 g/dL Platelet Count ≥ 100 x 109/L PT/INRa and PTT ≤ 1.3 x ULN Hepatic Total Bilirubinb ≤ 1.5 x ULN AST and ALT ≤ 2.5 x ULN Renal Serum Creatinine ≤ 1.5 mg/dL Abbreviations: ALT = alanine transaminase; ANC = absolute neutrophil count; AST = aspartate aminotransferase; INR = international normalized ratio; LLN = lower limit of normal; PT = prothrombin time; PTT = partial thromboplastin time; ULN = upper limit of normal.

   a Subjects receiving anticoagulation treatment may be allowed to participate with INR established within the therapeutic range prior to enrollment.

   b Subjects with known Gilbert's syndrome must have a total bilirubin < 3.0 x ULN).

   c If serum creatinine is > 1.5 mg/dL, calculate creatinine clearance using standard Cockcroft-Gault formula. Creatinine clearance must be ≥ 50 mL/min to be eligible.
6. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

1. Females who report they are pregnant or breast-feeding at the time of screening will not be eligible for this study. Female participants of child-bearing potential will have a urine pregnancy test prior to infusion of the study radiotracer to confirm they are not pregnant.
2. Patients who have any splenic disorders, or had splenectomy, that in the opinion of an investigator could compromise protocol objectives.
3. Inability to tolerate imaging procedures in the opinion of the investigator or treating physician.
4. Serious or unstable medical or psychological conditions that, in the opinion of the investigator would compromise the subject's safety or successful participation in the study.
5. Ineligible for the LIMIT Melanoma Trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Zirconium Zr 89 Crefmirlimab Berdoxa uptake | 21 days
  Zirconium Zr 89 Crefmirlimab Berdoxa measured uptake *(by standard uptake value) on Baseline and post-Treatment PET/CT scans in tumor lesions and lymphoid organs.
Change in uptake post therapy | 21 days
  Measurement of change in Zirconium Zr 89 Crefmirlimab Berdoxa uptake between Baseline and post-Treatment PET/CT scans in tumor lesions and lymphoid organs.

SECONDARY OUTCOMES:
Post therapy outcomes | until the end of the study, usually about 3 years
  Association between change in tumor Zirconium Zr 89 Crefmirlimab Berdoxa uptake and objective response, progression free survival, and overall survival.
CD8+ TIL density in tumor | 2 months
  Association between tumor Zirconium Zr 89 Crefmirlimab Berdoxa uptake and CD8+ TIL density in biopsied tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- Perleman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States